CLINICAL TRIAL: NCT05327699
Title: Glutamatergic Adaptation to Stress as a Mechanism for Anhedonia and Treatment Response With Ketamine
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Treadway, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00003476; R01MH126083-01A1 (NIH)
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
Keywords: Neuroscience; Stress response
MeSH Terms: conditions — Depressive Disorder, Major; Fractures, Stress | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Major depressive disorder (MDD) Ketamine (Experimental): Participants randomized to the ketamine arm will receive a single intravenous (IV) infusion of ketamine at 0.5mg/kg through an indwelling catheter over a 40-100min period.
  Interventions: Drug: Ketamine
- Major depressive disorder (MDD) Placebo (Placebo Comparator): Participants randomized to the placebo arm will receive a single intravenous (IV) infusion of saline through an indwelling catheter over a 40-100min period.
  Interventions: Other: Placebo
- Healthy Controls (No Intervention): The subjects in this group will not receive any intervention.

INTERVENTIONS:
Drug: Ketamine — A single intravenous (IV) infusion of ketamine calculated at 0.5mg/kg through an indwelling catheter over a 40-100min period.
  Other Names: Ketalar
  Arms: Major depressive disorder (MDD) Ketamine
Other: Placebo — A single intravenous (IV) infusion of saline through an indwelling catheter over a 40-100min period.
  Arms: Major depressive disorder (MDD) Placebo

SUMMARY:
The main purpose of this study is to investigate the effects of ketamine on decision-making and emotion processing in a sample of individuals diagnosed with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
The main purpose of this study is to understand the effects of sub-anesthetic ketamine doses on varying functional domains of depression such as anhedonia, decision-making, and emotion processing in subjects diagnosed with Major Depressive Disorder (MDD). The study will evaluate these effects using a combination of questionnaires, neuroimaging techniques, and behavioral tasks. The clinical trial portion will only include subjects with MDD (Major Depressive Disorder). A separate group of healthy controls, n=60, will be invited to only complete a behavioral/interview session and one neuroimaging session.The healthy controls group will not be randomized nor receive any study intervention and will only serve to collect performance baseline measures. The primary aims of this study are to evaluate 1) the glutamate stress response in MDD patients and matched controls by whole-brain imaging, 2) the multi-modal associations between glutamate stress response and neuroimaging and behavioral assessments of motivation and valuation, and 3) the effect of ketamine versus placebo on glutamate stress response in MDD subjects.

ELIGIBILITY:
Inclusion Criteria:

MDD Patients:

* willing and able to give written informed consent
* men or women, 18-65 years of age
* primary diagnosis of DSM-V MDD, current, as diagnosed by the SCID-I
* score of ≥20 on the Beck Depression Inventory, which will include patients characterized as having "moderate/severe" (20-28) or "very-severe" (29-63) depressive symptoms
* off all antidepressant therapy for at least 8 weeks prior to the baseline visit

Healthy Controls:

* willing and able to give written informed consent
* men or women, 18-65 years of age

Exclusion Criteria:

MDD Patients:

* history of any bipolar disorder or psychotic disorder
* active psychotic symptoms of any type
* substance abuse/dependence within 6 months of study entry (as determined by SCID)
* unstable cardiovascular, endocrinologic, hematologic, hepatic, renal, or neurologic disease (as determined by physical examination and laboratory testing), including upper respiratory disease or asthma, glaucoma or porphyria.
* active suicidal ideation as determined by a score ≥3 on the Columbia Suicide Severity Rating Scale (C-SSR)
* use of any recreational drugs as confirmed by urine drug screen at the time of scanning
* pregnancy or lactation
* use of glucocorticoids at any time during the study
* Raynaud's disease that may interfere with the cold-pressor
* contraindications for MRI
* MMSE score <28
* elevated blood pressure prior to infusion (systolic > 160 or diastolic >100)
* history of treatment resistance as determined by ATRQ
* prior adverse reaction to ketamine
* use of antipsychotic medications
* use of greater than 2mg daily of lorazepam or similar benzodiazipine.
* Regular smoker as self-reported

Healthy Controls:

* evidence of any psychiatric disorder with exception of specific phobia, and no history of any psychiatric disorder except mild past substance use disorder as diagnosed by the SCID-I
* history of any substance abuse within the last 6 months
* use of any recreational drugs as confirmed by urine drug screen at the time of scanning
* pregnancy or lactation
* use of glucocorticoids at any time during the study
* Raynaud's disease that may interfere with the cold-pressor
* contraindications for MRI
* MMSE score <28
* Regular smoker as self-reported

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in glutamate concentration in the medial prefrontal cortex (mPFC) | Baseline, 24 hours post-infusion, 14 days post-infusion
  The glutamate concentration in the mPFC as determined by in vivo magnetic resonance spectroscopy (MRS) at a field strength of 3 Tesla (3T) using standard MRS protocols. The levels of glutamate metabolite will be quantified using a custom quantification algorithm for modelling the background noise inherent in NMR (Nuclear Magnetic Resonance) signals. In MDD participants receiving ketamine, acute stress challenges will result in decreased glutamate in mPFC at 24 hrs that will be sustained at 2 weeks.

OTHER OUTCOMES:
Change in Apathy Motivation Index (AMI) | Baseline, 24 hours post-infusion, 14 days post-infusion
  The AMI is an 18-item self-report index of apathy and motivation. It is used to assess the different mechanisms of sub-clinical lack of motivation. It covers motivation within three dissociable domains: cognitive, emotional/affective and behavioral. Every domain contains 6 items that is each scored from 0-4, with a higher mean score indicating greater apathy.
Change in Motivation and Pleasure Scale (MAP-SR) | Baseline, 24 hours post-infusion, 14 days post-infusion
  The mood and pleasure questionnaire is a 15-item self-report measure of severity of negative symptoms. This scale will be used to assess self-reported changes in motivational anhedonic symptoms. All items are rated on a 5-point Likert scale; higher scores reflect greater pathology. .
Change in Dysfunctional Attitudes Scale - Short Form (DAS-SF) | Baseline, 24 hours post-infusion, 14 days post-infusion
  The DAS-SF is a self-report questionnaire containing nine items and utilizes an item-response analysis to provide an efficient and accurate assessment of dysfunctional attitudes. Subjects will rate their agreement to each of the 9 statements on a Likert scale of agreement from 1 to 5. Scores could range from 9 to 45, with higher scores reflecting more dysfunctional attitudes.
Change in Perceived Stress Scale (PSS) | Baseline, 24 hours post-infusion, 14 days post-infusion
  The Perceived Stress Scale (PSS) is a psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  Scores ranging from 0-13 would be considered low stress, 14-26 would be considered moderate stress and 27-40 would be considered high perceived stress.
Change in State-Trait Anxiety Inventory (STAI) | Baseline, 24 hours post-infusion, 14 days post-infusion
  The State-Trait Anxiety Inventory (STAI) is used measure trait and state anxiety. It consists of 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater levels of anxiety.
Change in Mini-Mental State Exam (MMSE) | Baseline, 24 hours post-infusion, 14 days post-infusion
  The MMSE is a 30-item interviewer-administered questionnaire widely used for the evaluation of general cognitive functioning and identification of altered mental status. A score ≤24, indicates evidence of more than mild cognitive impairment.
Change in Reaction Time Task (RTT) | Baseline, 24 hours post-infusion, 14 days post-infusion
  The RTT provides measures of simple and choice movement and reaction time tasks and is divided into 5 stages requiring increasingly complex chains of responses and providing distinction between reaction (or decision) time and movement latencies. Reaction times are typically 0.2 seconds (s) to 0.9 s. Shorter reaction times indicate better cognitive processes of perception and response execution.
Change in Reinforcement Learning Task | Baseline, 24 hours post-infusion, 14 days post-infusion
  Participants will be asked to perform three runs of an instrumental learning task. For each run, one pair of visual stimuli will be randomly presented, with one stimulus above and one below a fixation cross (counterbalanced). The subject will be instructed to choose the upper or lower stimulus by pressing one of two keys. After 4 seconds, the choice will be circled in red and the outcome (either "Nothing", "Gain", "Loss" or "Look") will be presented, accompanied by the image of a $1 bill in the event of gain, loss and look outcomes. In sum, to win money the subjects will have to learn, by trial and error, the stimulus-outcome associations. Higher stimulus-outcome associations made will indicate increased cognitive function.
Change in Apathy Evaluation Scale (AES) | Baseline, 24 hours post-infusion, 14 days post-infusion
  The AES addresses characteristics of goal directed behavior that reflects apathy including behavioral, cognitive and emotional indicators. It consists of 18 items; Items are scored on 4-point Likert scale with descriptors for the "self" version (not at all true, slightly true, somewhat true, very true). The score range for the complete AES (total AES score) is 18 to 72, with a lower score indicating greater apathy.
Change in UCLA Loneliness Scale | Baseline, 24 hours post-infusion, 14 days post-infusion
  The UCLA (University of California, Los Angeles) Loneliness Scale is a 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item on a scale from 1 (Never) to 4 (Often). Higher scores indicate higher levels of feeling lonely or isolated.
Change in Digit Symbol Task (DST) | Baseline, 24 hours post-infusion, 14 days post-infusion
  The Digit Symbol Task consists of rows of blank squares, each printed with a randomly assigned number. The test involves graphomotor speed, visual scanning and memory, with about half of the variance being accounted for by graphomotor speed, a third by visual scanning and 4-5% by memory. Scores range from 0 to 100. Higher scores indicate higher cognitive function.
Change in Finger Tapping Task (FTT) | Baseline, 24 hours post-infusion, 14 days post-infusion
  This task uses a specially adapted tapper that the subject taps as fast as possible using the index finger. The subject is given 5 consecutive 10-second trials for the preferred and non-preferred hands. The finger tapping score is the mean of 5 trials and is computed for each hand. Lower scores indicate higher levels of brain dysfunction and higher scores are indicative of better brain function.
Change in Effort-Based Decision-Making Task | Baseline, 24 hours post-infusion, 14 days post-infusion
  This task will require subjects to make repeated choices between an effortful option and a no-effort option. The effortful option varies in the amount of effort required (20%, 50%, 80% and 100% of the subject's individually-calibrated maximum effort, set for each individual prior to scan), measured in speeded button presses. The reward magnitude for the no-effort option remains constant ($1.00), while the reward magnitude for the high-effort option ranges from $1.00 to $5.00. These tasks assess how much effort a person is willing to exert for a given level of reward. Higher reward scores indicate a higher input of effort.
Change in Effort-Discounting Task | Baseline, 24 hours post-infusion, 14 days post-infusion
  In this task, subjects will first be asked to make a series of speeded button presses to calibrate in their rates of effortful responding. Subjects will be given three trial task choices where they will be asked to push a button as quickly as possible for a total of 20 seconds. Based on the average maximum speed, subjects will then be presented with choices between performing 100%, 80%, 50%, and 20% of this effort in exchange for various amounts of money ($1.00-$5.00), and doing nothing to win $1.00. The number of participants opting for the higher choice of reward will be recorded.
Change in MoVER Task - Navigate | Baseline, 24 hours post-infusion, 14 days post-infusion
  In this task, subjects will be trained on different computerized mazes with varying difficulties/lengths. There will be a group of easy mazes and a group of hard mazes. After a subject has sufficiently learned the mazes (defined as reaching the end of a maze by a specified goal time), he or she will begin the task itself. In this task, subjects will be exposed to "navigate" trial tasks. In "navigate" trials, subjects will have to reach the end of the maze for a varying known or unknown reward amount (ranging from $0-10). The number of participants who complete the task will be recorded.
Change in MoVER Task- Passive Viewing | Baseline, 24 hours post-infusion, 14 days post-infusion
  In this task, subjects will be trained on different computerized mazes with varying difficulties/lengths. There will be a group of easy mazes and a group of hard mazes. After a subject has sufficiently learned the mazes (defined as reaching the end of a maze by a specified goal time), he or she will begin the task itself. In this task, subjects will be exposed to "passive viewing" trials, subjects will watch as they are navigated through the maze without needing to actively respond or move. The number of participants who complete the task will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Treadway, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All members of this research team are strongly committed to open access data policies and the dissemination of research results in a timely manner. The results of the study will be published in a timely manner in the most appropriate journals and presented at relevant national and international conferences. Data will include participant data that underlie the results reported in a given article, after deidentification. No other documents will be included.
Time Frame: Data will be available within 1 year after completion of the grant.
Access Criteria: Data will be shared via NDAR (National Database for Autism Research). Data will be available within 1 year after completion of the grant. Investigators will need to access data via NDAR.Data can be used for any purpose that NDAR approves.